CLINICAL TRIAL: NCT07174401
Title: Rocklatan Trial With Optical Coherence Tomography Study of Retinal Perfusion
Brief Title: Rocklatan Retinal Perfusion OCT Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, David Huang, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU IRB0029104
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
Keywords: Glaucoma; Rocklatan
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator will assign one eye to use the study drug, while the other eye (control) will remain on the clinically prescribed medication. The identity of the eye drop will be masked to both participants and study personnel who perform testing procedures or data analysis. The university research pharmacy will provide label masked bottles for each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Eye with Diagnosed Glaucoma (Experimental)
  Interventions: Drug: Rocklatan eye drops will be instilled nightly in one eye diagnosed with glaucoma for up to 12 months.; Device: Two optical coherence tomography (OCT) devices will be used to assess blood flow changes.
- Control Eye (No Intervention): This is also an eye with glaucoma, but the control eye will use clinically prescribed medication instead of the study drug.

INTERVENTIONS:
Drug: Rocklatan eye drops will be instilled nightly in one eye diagnosed with glaucoma for up to 12 months. — The eye not selected as the study eye will be used for comparison so both eyes will be imaged with the study devices to assess blood flow changes.
  Arms: Eye with Diagnosed Glaucoma
Device: Two optical coherence tomography (OCT) devices will be used to assess blood flow changes. — One OCT device is FDA-cleared while the other is still experimental. Both devices assess blood flow in different ways.
  Arms: Eye with Diagnosed Glaucoma

SUMMARY:
The main purpose of this study is to learn more about how Rocklatan eye drops affects blood flow in the eye. The secondary purpose is to see if our study devices can detect changes in blood flow before and after instillation of Rocklatan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with both eyes with open angle glaucoma.
2. Abnormal VF (glaucomatous pattern with PSD abnormal at p<0.05 or GHT outside normal limits) on most recent two clinic visits on chart review
3. Glaucomatous disc abnormality on chart review and confirmed on baseline disc photograph
4. Overall average NFL thickness > 55 μm measured by Heidelberg Spectralis OCT -Glaucoma Module Premium Edition (chart review), consistent with early glaucoma
5. NFLP-CD deficit (below 5 percentile of normal) in any of the 8 sectors on the initial baseline visit
6. The difference in baseline NFLP-CD between the left and right eye should be less than 5% (% of area).
7. IOP >= 17 mm Hg on the most recent two clinic visits (chart review) after monotherapy with latanoprost in both eyes.

Exclusion Criteria:

1. Best corrected visual acuity worse than 20/30 on chart review of most recent clinic visit
2. Age < 21 years at baseline
3. Eye disease that could affect VF, NFL thickness, or NFLP (e.g., visually significant cataract, AMD, diabetic retinopathy, and optic neuropathy) at any study visit
4. OCT and OCTA scans not meeting quality criteria at baseline
5. Inability to cooperate with study procedures
6. Inability to commit to the study visits

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Nerve Fiber Layer Plexus Capillary Density (NFLP CD) | From enrollment to end of treatment at 11-12 months
  The primary outcome measure will be change in the overall peripapillary NFLP CD measured at 6 months and 11-12 month endpoint visits compared to baseline values.

SECONDARY OUTCOMES:
Total Retinal Blood Flow (TRBF) | From enrollment to end of treatment at 11-12 months
  Secondary outcome measures will include change in the TRBF measured at 6 months or 11-12 month endpoint visits compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute - Oregon Health & Science University, Portland, Oregon, United States